CLINICAL TRIAL: NCT04569942
Title: Australasian Resuscitation In Sepsis Evaluation: FLUid or Vasopressors In Emergency Department Sepsis
Acronym: ARISE FLUIDS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANZIC-RC/SP002
Record Dates: First submitted 2020-09-23; First posted 2020-09-30 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Shock, Septic
Keywords: septic shock; vasopressor; Resuscitation Fluids
MeSH Terms: conditions — Shock, Septic | interventions — Vasoconstrictor Agents; Fluid Therapy

STUDY DESIGN:
Intervention Model Description: randomized, controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vasopressor (Active Comparator): a restricted fluids and early vasopressor strategy
  Interventions: Drug: Vasopressor
- Fluids (Active Comparator): a larger intravenous (IV) fluid volume and later vasopressor strategy
  Interventions: Other: Fluids

INTERVENTIONS:
Drug: Vasopressor — Cease IV fluid resuscitation. If persisting hypotension and/or hypoperfusion commence a vasopressor infusion (e.g. noradrenaline) and titrate according to local practice to achieve target MAP. The target MAP will be determined by the treating clinician. Reassess at least hourly for up to 6 hours post-randomisation, then as clinically required in conjunction with the protocol. Boluses of 250ml of IV fluids are permitted if deemed indicated by the treating clinician.
  Arms: Vasopressor
Other: Fluids — An fluid bolus of up to 1000ml will be administered over a maximum of 1 hour, if required, for persisting hypotension and/or hypoperfusion. Reassess at least hourly to 6 hours post-randomisation, then as clinically required in conjunction with the protocol. Further IV fluid boluses of 500ml are recommended as clinically indicated to achieve the target MAP. The target MAP will be determined by the treating clinician. Haemodynamic resuscitation will be guided by usual clinical assessment including vital signs, mentation, perfusion, and urine output until the treating clinician determines fluid resuscitation is no longer clinically required. A minimum of 2-3 L (30 ml/kg), including pre-randomisation fluids, is recommended within 3 hours of ED arrival consistent with the SSC guidelines, unless clinically contraindicated. Vasopressors may be commenced if blood pressure remains below target despite optimal fluid resuscitation as determined by the treating clinician.
  Arms: Fluids

SUMMARY:
This multicentre, randomised controlled trial will enrol 1000 patients presenting with septic shock to the emergency department (ED) of participating hospitals in Australia and New Zealand. Participants will receive haemodynamic resuscitation with either a restricted fluids and early vasopressor regimen or a larger initial IV fluid volume with later introduction of vasopressors if required. Clinical care including the type of resuscitation fluid and vasopressor agent, will otherwise be in accordance with accepted standard care and according to clinician discretion. The study intervention will be delivered for at least 6 hours and up to 24 hours post-randomisation. Participants will be followed for up to 12 months and outcomes analysed on an intention-to-treat basis.

DETAILED DESCRIPTION:
The ARISE FLUIDS study is a multicentre, randomised, parallel group clinical trial of a restricted fluids and early vasopressor strategy compared to a larger initial IV fluid volume and later vasopressors for the haemodynamic resuscitation of patients with septic shock presenting to the ED. It will be conducted in hospitals in Australia and New Zealand with 1000 patients recruited over a 3-year period.

Each patient meeting all of the inclusion and none of the exclusion criteria will be randomised to receive haemodynamic resuscitation using either a restricted fluid and early vasopressor regimen (vasopressors arm) or a larger initial fluid resuscitation volume (fluids arm) followed by later introduction of vasopressors (if required). The intervention will be commenced in the ED and delivered for at least 6 hours, and up to 24 hours post-randomisation if admitted to the ICU or other critical care area where the study protocol can be faithfully delivered. Treatment will revert to usual care as determined by the treating clinician when the patient is transferred to a non-critical care ward. All enrolled participants will be followed up and assessed for the defined study outcomes.

Participants will be identified using a systematic approach to screening and assessment of patients with possible sepsis presenting to the ED in accordance with standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Clinically suspected infection;
* Systolic blood pressure (SBP) <90 mm Hg or mean arterial pressure (MAP) <65 mm Hg, despite a ⩾1000ml cumulative total bolus of IV fluid administered over a maximum of 60 minutes; including pre-hospital boluses;
* Arterial or venous blood lactate >2.0 mmol/L;
* At least one dose of an intravenous antimicrobial has been commenced.

Exclusion Criteria:

* Age <18 years;
* Confirmed or suspected pregnancy;
* Transferred from another acute care facility;
* Hypotension suspected to be due to a non-sepsis cause;
* >2L total IV fluid administered (including prehospital fluids but excluding drugs and flushes);
* More than 6 hours has elapsed since presentation to the ED or more than 2 hours has elapsed since last inclusion criterion has been met;
* Treating clinician considers that one or both of the treatment regimens are not suitable for the patient or the study protocol cannot be delivered e.g. limitation of care, requirement for immediate surgery;
* Death is considered imminent or inevitable;
* Underlying disease that makes survival to 90 days unlikely;
* Inability to follow patient up to day-90 e.g. unstable accommodation, overseas visitor;
* Previously enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-11-03 (Estimated)

PRIMARY OUTCOMES:
Days alive and out of hospital | From randomisation until 90 days post- randomization
  the number of days alive and out of hospital at 90 days post randomization

SECONDARY OUTCOMES:
Mortality | From randomisation until 90 days post- randomization
  All-cause mortality
Time from randomization until death | From randomisation until 90 days post- randomization
  Time from randomization until death
Days alive and at home | From randomisation until 90 days post- randomization
  Days alive and at home at 90 days post-randomisation
Ventilator-free days to day 28 | From randomisation until 28 days post- randomization
  Number of days not on invasive mechanical ventilation
Vasopressor-free days to day 28 | From randomisation until 28 days post- randomization
  Number of days not on vasopressors
Renal replacement therapy-free days to day 28 | From randomisation until 28 days post- randomization
  Number of days not on renal replacement therapy
Death or disability at 6 months | at 6 months post randomization
  Death or disability as measured by the World Health Organization Disability Assessment Schedule (WHODAS)
Death or disability at 12 months | at 12 months post randomization
  Death or disability as measured by the World Health Organization Disability Assessment Schedule (WHODAS)

OTHER OUTCOMES:
Incidence of invasive mechanical ventilation | From randomisation until 90 days post- randomization
  Incidence of invasive mechanical ventilation
Duration of invasive mechanical ventilation | From randomisation until 90 days post- randomization
  Duration of invasive mechanical ventilation
Incidence of acute renal replacement therapy | From randomisation until 90 days post- randomization
  Incidence of acute renal replacement therapy
Duration of acute renal replacement therapy | From randomisation until 90 days post- randomization
  Duration of acute renal replacement therapy
Incidence of vasopressor support | From randomisation until 90 days post- randomization
  Incidence of vasopressor support
Duration of vasopressor support | From randomisation until 90 days post- randomization
  Duration of vasopressor support
Emergency Department length of stay | From randomisation until 90 days post- randomization
  Emergency Department length of stay
Intensive care unit length of stay | From randomisation until 90 days post- randomization
  Intensive care unit length of stay
Hospital length of stay | From randomisation until 90 days post- randomization
  Hospital length of stay
In hospital mortality | From randomisation until 90 days post- randomization
  Patients who die in hospital
Mortality at 6 months | 6 Months post- randomization
  mortality at 6 months
Mortality at 12 months | 1 year post- randomization
  mortality at 12 months
Quality of life at 6 months | 6 months post- randomization
  Patient quality of life as measured by the EuroQol Group 5 dimensions 5 levels survey (EQ-5D-5L)
Quality of life at 12 months | 1 year post- randomization
  Patient quality of life as measured by the EuroQol Group 5 dimensions 5 levels survey (EQ-5D-5L)
Cost-effectiveness measured as cost/quality-adjusted life year (QALY) | 1 year post- randomization
  cost effectiveness measured as cost per quality-adjusted life year

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Peake, MBBS, Study Chair — Monash University
Locations (50):
- Australia (44):
  - Bankstown Hospital, Bankstown, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Nepean Hosital, Kingswood, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - Royal North Shore Hosptial, Sydney, New South Wales
  - Ryde Hospital, Sydney, New South Wales
  - Tamworth Hospital, Tamworth, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Darwin & Palmerston Hospital, Darwin, Northern Territory
  - The Prince Charles Hospital, Brisbane, Queensland
  - QE II Jubilee Hospital, Brisbane, Queensland
  - Bundaberg Hospital, Bundaberg, Queensland
  - Caboolture Hospital, Caboolture, Queensland
  - Cairns Hospital, Cairns, Queensland
  - Hervey Bay Hospital, Hervey Bay, Queensland
  - Ipswich Hospital, Ipswich, Queensland
  - Mackay Base Hospital, Mackay, Queensland
  - Robina Hospital, Robina, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Sunshine Coast university hospital, Sunshine Coast, Queensland
  - Toowoomba Hospital, Toowoomba, Queensland
  - Townsville Hospital, Townsville, Queensland
  - The Queen Elizabeth Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Streaky Bay, South Australia
  - Ballarat Base Hospital, Ballarat, Victoria
  - Bendigo Hospital, Bendigo, Victoria
  - Casey Hospital, Berwick, Victoria
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Dandenong Hospital, Dandenong, Victoria
  - Northern Hospital, Epping, Victoria
  - Angliss Hospital, Ferntree Gully, Victoria
  - St. Vincent's Hospital, Fitzroy, Victoria
  - Barwon Health Geelong Hospital, Geelong, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Maroondah Hospital, Ringwood East, Victoria
  - Wangaratta Hospital, Wangaratta, Victoria
  - Bunbury Hospital, Bunbury, Western Australia
  - St John of God Hospital, Midland, Western Australia
  - St John of God Murdoch Hospital, Murdoch, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
  - Fiona Stanley Hospital, Perth, Western Australia
- St. Vincent's University Hospital, Elm Park, Dublin, Ireland
- New Zealand (5):
  - Auckland City Hospital, Auckland, North Island
  - Dunedin Hospital, Dunedin, Otago
  - Middlemore Hospital, Middlemore, Otahuhu
  - Taranki Hospital, Hawera
  - Wellington Hospital, Wellington

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be available one year after the publication date for a 2 year period
Access Criteria: Data requests can be submitted to the ARISE FLUIDS Management Committee, via the project manager, Ms Belinda Howe, at belinda.howe@monash.edu. The data will be made available following the submission of an appropriate research question, approval of the application by the ARISE FLUIDS management committee, and execution of a data sharing agreement.
URL: https://www.monash.edu/medicine/sphpm/anzicrc

REFERENCES:
- [Derived] Howe BD, Macdonald SPJ, Arendts G, Bellomo R, Burcham J, Delaney A, Egerton-Warburton D, Fatovich D, Fraser JF, Higgins A, Jones P, Keijzers G, Milford E, Udy AA, Williams P, Young P, Peake SL. Australasian Resuscitation In Sepsis Evaluation: FLUid or vasopressors In emergency Department Sepsis (ARISE FLUIDS) trial: study protocol. BMJ Open. 2025 Jul 20;15(7):e101215. doi: 10.1136/bmjopen-2025-101215. PMID 40685240
- See also: SAP for trial — https://www.monash.edu/medicine/sphpm/anzicrc/research/protocols-saps